CLINICAL TRIAL: NCT05911438
Title: Accelerated Recovery for Total Knee Replacement Surgery With Preoperative Intravenous Iron Combined With Human Erythropoietin for Rapid Hematopoietic Mobilization to Prevent Postoperative Anemia: a Multicenter Randomized Controlled Study
Brief Title: Accelerated Recovery for Total Knee Replacement Surgery With Preoperative Intravenous Iron Combined With Human Erythropoietin for Rapid Hematopoietic Mobilization to Prevent Postoperative Anemia
Acronym: Hematoboost
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Fuxing Pei, Director of Department of Orthopaedic Surgery, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HX-TKA-IV-001
Record Dates: First submitted 2023-06-09; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Total Knee Arthroplasty
Keywords: Human Erythropoietin; Ferric Derisomaltose Injection
MeSH Terms: interventions — ferric derisomaltose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Ferric Derisomaltose Injection (Monoferric) and Human Erythropoietin Injection (EPIAO); Other: Basic Treatment
- Control group (Placebo Comparator)
  Interventions: Other: Basic Treatment

INTERVENTIONS:
Drug: Ferric Derisomaltose Injection (Monoferric) and Human Erythropoietin Injection (EPIAO) — Ferric Derisomaltose Injection (Monoferric): 1000 mg, intravenous infusion 6±2 days before surgery; Human Erythropoietin Injection (EPIAO): 36000 IU, subcutaneous injection 6±2 days before surgery and 3±1 days after surgery.
  Arms: Experimental group
Other: Basic Treatment — Daily energy intake of 20-30 kcal/kg, with fat accounting for 20-30% of total energy; Iron: ≥15 mg/d, protein intake of 1.2-1.5 g/kg/d; Simultaneously enhance functional exercises.

SUMMARY:
This study is a randomized, placebo-controlled, multicenter research design to investigate the effectiveness and safety of a single-dose intravenous iron combined with HuEPO hematopoietic mobilization before surgery in patients undergoing unilateral total knee arthroplasty for the first time.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, multicenter research design to investigate the effectiveness and safety of a single-dose intravenous iron combined with HuEPO hematopoietic mobilization before surgery in patients undergoing unilateral total knee arthroplasty for the first time.

The study consists of a pilot trial and a formal trial. The pilot trial plans to enroll 20 subjects, with 10 subjects randomly assigned to the experimental group and 10 subjects to the control group. After the successful completion of the pilot trial, its safety and effectiveness, as determined by the investigators, hematologists, orthopedic surgeons, and statisticians, and the formal trial will be initiated. The relevant information and results will also be submitted to the ethics review committee. The formal trial plans to enroll 399 eligible subjects, with a random allocation ratio of 2:1 to the experimental group or the control group.

To ensure the safety of the subjects, the last subject in the pilot trial will be followed up for 21 days after surgery. The safety and effectiveness of the pilot trial results will be discussed by the investigators, hematologists, orthopedic surgeons, and statisticians before initiating the formal trial. The timing of medication, sample size, and visit points in the formal trial may be adjusted appropriately based on the results of the pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years (inclusive) and no gender restriction at the time of signing the informed consent form (ICF).
* Patients who meet the diagnostic criteria for osteoarthritis according to the American College of Rheumatology (ACR) and are undergoing primary total knee arthroplasty due to end-stage osteoarthritis. Flexion deformity <30°, varus deformity <30°, valgus deformity <20°.
* Baseline hemoglobin level: 100g/L < Hb < 130g/L.
* No deep venous thrombosis observed on preoperative bilateral lower limb venous color Doppler ultrasound.
* The subject understands and voluntarily signs the written informed consent form (ICF) and is capable of complying with the scheduled visits and related procedures as outlined in the protocol.

Exclusion Criteria:

* Known allergy to any excipients in the investigational drugs iron sucrose and erythropoietin or a history of multiple allergies.
* Mean corpuscular volume (MCV) > 100 fL.
* Numeric Rating Scale (NRS) score ≥ 3.
* Presence of iron overload (serum ferritin > 800 ng/ml) or iron utilization disorders (such as hemochromatosis and iron deposition disorders).
* Blood disorders other than iron-deficiency anemia.
* Blood transfusion within the past 30 days.
* Use of iron preparations or HuEPO for the treatment of anemia within the past 30 days.
* History of deep vein thrombosis or pulmonary embolism.
* Patients with hypophosphatemia due to various causes.
* BMI < 18.5 kg/m2 or body weight < 50 kg.
* History of recent myocardial infarction, angina pectoris, cerebral infarction, or epileptic seizures within the past 6 months.
* Use of medications affecting coagulation and antiplatelet function within the past week.
* Moderate liver impairment: Decompensated liver cirrhosis or hepatitis, ALT, AST > 3 times the upper limit of normal (ULN).
* Moderate renal impairment: Serum creatinine (Cr) > 150 µmol/L.
* HIV or syphilis patients.
* Pregnant or lactating women.
* Participants who have previously participated in other clinical trials, provided the previous investigational drug exposure did not exceed 5 half-lives.
* Acute infection, rheumatoid arthritis, or significant joint inflammation.
* Patients deemed unsuitable to participate in this clinical trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin concentration | postoperative 14±3 days
  Hemoglobin concentration

SECONDARY OUTCOMES:
Total blood loss | postoperative 3±1 days
  Total blood loss
Transfusion rate and amount | postoperative 14±3 days
  Transfusion rate and amount
Assess changes in serum ferritin and transferrin saturation | postoperative 14±3 days and 28±5 days
  Assess changes in serum ferritin and transferrin saturation
Quality of life indicators (SF-12) | postoperative 28±5 days and 90±12 days
  Quality of life indicators (SF-12)
The rates of adverse events (AE) | postoperative 90±12 days
  Assessed according to NCI-CTCAE v5.0 criteria
The rates of serious adverse events (SAE) | postoperative 90±12 days
  Assessed according to NCI-CTCAE v5.0 criteria
The rates of laboratory abnormalities | postoperative 90±12 days
  Assessed according to NCI-CTCAE v5.0 criteria
The rates of adverse events leading to drug discontinuation | postoperative 90±12 days
  The rates of adverse events leading to drug discontinuation
The rates of adverse events leading to permanent discontinuation | postoperative 90±12 days
  The rates of adverse events leading to permanent discontinuation
The rates of adverse events leading to early withdrawal from the study | postoperative 90±12 days
  The rates of adverse events leading to early withdrawal from the study

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China